CLINICAL TRIAL: NCT03125512
Title: Comparing a Convenient Positional Therapy Device to CPAP for Treatment of Positional Obstructive Sleep Apnea, A Crossover Randomized Controlled Trial
Brief Title: Positional Therapy Versus CPAP for Positional OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OSA_RCT
Record Dates: First submitted 2017-04-09; First posted 2017-04-24 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea Syndromes; Positional sleep apnea; CPAP; Night Shift
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: 8-week randomized crossover trial with a 1 week washout period.
Who Masked: Outcomes Assessor
Masking Description: Research staff assessing the outcomes of the study, the scoring of the sleep studies, and data analyses will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Night Shift positional device (Experimental): Randomized to Night shift positional therapy first for 8 weeks, followed by CPAP for 8 weeks, with a 1 week washout period.
  Interventions: Device: Night Shift positional device
- Continuous positive airway pressure (Active Comparator): Randomized to CPAP first for 8 weeks, followed by positional therapy for 8 weeks, with a 1 week washout period.
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: Night Shift positional device — Night Shift is a small, positional therapy device that is worn at the back of the neck using a latex free silicone rubber strap. The strap is adjustable and is secured with a magnetic clasp. When a supine position is detected, the device vibrates with increasing intensity till the subject changes to a non-supine position.
  Arms: Night Shift positional device
Device: continuous positive airway pressure — Automated adjusting continuous positive airway pressure
  Arms: Continuous positive airway pressure

SUMMARY:
This is a crossover randomized controlled trial comparing a convenient positional therapy (PT) device to continuous positive airway pressure (CPAP) in the treatment of positional obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
This study aims to compare a convenient positional therapy (PT) device used for 8 weeks to continuous positive airway pressure (CPAP) used for 8 weeks in patients with positional obstructive sleep apnea (OSA) in a crossover randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and above
2. Epworth sleepiness scale 10 to 16
3. No CPAP treatment or PT treatment for past 6 months
4. A diagnosis of positional OSA based on a full in-laboratory overnight polysomnography with

   1. Total apnea/hypopnea index (AHI) >10 /hour and non-supine AHI < 10/hour
   2. Supine AHI greater than or equal to two times the non-supine AHI
   3. At least 15 minutes of supine and non-supine sleep

Exclusion Criteria:

1. Epworth sleepiness scale ≥17
2. Commercial driving
3. Unable or unwilling to use both treatments (CPAP and PT)
4. Concurrent use of therapy for OSA such as mandibular advancement splints
5. Conditions that preclude the ability to lie in a non-supine position, for example a shoulder injury
6. Uncontrolled severe medical/psychiatric conditions such as severe chronic heart failure, malignancy.
7. Patients with pacemaker
8. Skin sensitivity around the neck and/or open wound around their neck

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale ( ESS) | 8 weeks after the beginning of each intervention
  Difference in sleepiness ( PT minus CPAP) measured by the Epworth Sleepiness Scale ( ESS) after 8 weeks of device use

SECONDARY OUTCOMES:
Functional Outcomes of Sleep Questionnaire ( FOSQ) | 8 weeks after the beginning of each intervention
  Difference in FOSQ
36-Item Short Form Survey (SF-36) | 8 weeks after the beginning of each intervention
  Difference in SF-36
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks after the beginning of each intervention
  Difference in PSQI
Apnea-hypopnea Index ( AHI, events/hr) | 8 weeks after the beginning of each intervention
  Difference in AHI
DASS21 questionnaire | 8 weeks after the beginning of each intervention
  Difference in mood symptoms ( DASS21)
Patient adherence ( hours of device use per night) | 8 weeks after the beginning of each intervention
  Compare patient adherence based on device download information
Patient preference | Upon study completion at week 17
  patient preference for treatment modality will be assessed via a questionnaire
Oxygen desaturation index (3%) and lowest oxygen saturation ( %) | 8 weeks after the beginning of each intervention
  Oxygen indices

CONTACTS AND LOCATIONS:
Overall Officials: Yingjuan Mok, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mok Y, Tan A, Hsu PP, Seow A, Chan YH, Wong HS, Poh Y, Wong KKH. Comparing treatment effects of a convenient vibratory positional device to CPAP in positional OSA: a crossover randomised controlled trial. Thorax. 2020 Apr;75(4):331-337. doi: 10.1136/thoraxjnl-2019-213547. Epub 2020 Jan 2. PMID 31896735